CLINICAL TRIAL: NCT03213158
Title: Ixazomib for Desensitization in Kidney Transplantation
Brief Title: Ixazomib for Desensitization
Acronym: IXADES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0429; A534280 (Other: UW Madison); SMPH\MEDICINE\NEPHROLOGY (Other: UW Madison); Protocol ver 3June 2019 (Other: HS-IRB UW, Madison)
Record Dates: First submitted 2017-04-26; First posted 2017-07-11 (Actual); Results first posted 2022-05-11 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Kidney Diseases; End Stage Renal Disease
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Highly sensitized kidney transplant candidates (Experimental): The study population will include all highly sensitized kidney transplant candidates on the waitlist for more than 24 months at University of Wisconsin.
  Interventions: Drug: Ixazomib Oral Capsule

INTERVENTIONS:
Drug: Ixazomib Oral Capsule — Highly sensitized kidney transplant candidates on the waitlist for more than 24 months will receive ixazomib 3 mg (and dexamethasone 20 mg) on days 1, 8, and 15 of a 28 cycle. Patients will take ixazomib and dexamethasone for twelve (12) 28-day cycles.

SUMMARY:
The purpose of this research study is to find out how well ixazomib (the study drug) works to desensitize highly sensitized kidney transplant recipients.

DETAILED DESCRIPTION:
This is a pilot exploratory, proof of concept, open-label, single-center phase II investigator initiated clinical trial entitled IXAzomib for DESensitization (IXADES). The purpose of the study is (1) to examine the safety and efficacy of ixazomib for desensitization of highly sensitized kidney transplant candidates and (2) to conduct mechanistic studies to address the role of HLA and non-HLA antibodies, T and B cell phenotypes, and BAFF/APRIL in immune monitoring of sensitized kidney transplant candidates.

Specific Aim 1. To determine the safety and efficacy of ixazomib as a desensitization strategy. There is currently no effective desensitization strategy for highly sensitized patients defined as calculated Panel of Reactive Antibodies (cPRA) ≥ 80%. For this study, 10 highly sensitized kidney transplant candidates on the waitlist for more than 24 months will receive ixazomib 3 mg (and dexamethasone 20 mg) on days 1, 8, and 15 of a 28 cycle for 12 months. The primary objective is to evaluate the safety (distal neuropathy, thrombocytopenia, and gastrointestinal symptoms) and efficacy (decline in cPRA > 20%) of ixazomib. The secondary efficacy endpoint is transplantation rate within 12 months of therapy.

Specific Aim 2. Identify immune indices which predict the course of disease and/or response to treatment in highly sensitized patients. Mechanistic studies will use bone marrow and blood obtained from subjects in Aim 1 to determine the effect of treatment on immune regulation and reconstitution after therapy. Since the bone marrow microenvironment produces BAFF/APRIL and supports plasma cell maturation,the effect of therapy on the generation of BAFF/APRIL will be determined by bone marrow mesenchymal stem cells and the survival of bone marrow-derived plasma cells after desensitization. Specifically it's proposed to:

* Identify if bone marrow plasma cells, IgG subsets, and levels including free light chains, and circulating BAFF/APRIL predict outcomes.
* Determine if treatment is effective in downregulating circulating BAFF/APRIL and anti-HLA, endothelin-1 type A receptor (ETAR), angiotensin type 1 receptor (AT1R), and complement fixing C1q antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18-70 years of age.
* Able to provide informed consent.
* Female patients who are postmenopausal for at least 1 year before the screening visit, or are surgically sterile, or If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 30 days after the last dose of study drug, OR agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following: Agree to practice effective barrier contraception during the entire study treatment period and through 30 days after the last dose of study drug, or Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Patients must be highly sensitized with a cPRA ≥ 80%
* Be active on the waitlist for kidney transplantation > 24 months to confirm their inability to receive a deceased donor transplant because of their sensitization status.
* Patients must meet the following clinical laboratory criteria:

  1. Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet count ≥ 75,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
  2. Hemoglobin higher than 6 g/dL
  3. Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN).
  4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Major surgery requiring hospitalization within 6 months before enrollment
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Inability to take oral medication
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Grade 2 or greater peripheral neuropathy according to NCI Common Terminology Criteria for Adverse Events (CTCAE)
* Participation in other interventional clinical trials, including those with other investigational agents not included in this trial, within 6 months of the start of this trial and throughout the duration of this trial
* Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not
* Active or treated infection for HIV, HCV or HBV
* History of Liver cirrhosis, biopsy confirmed
* Elevated transaminases (greater than 3 times the upper limit of normal)
* Known hypersensitivity to ixazomib
* Active substance abuse by self-report or medical record

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arjang Djamali, MD, MS, FASN, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Wilson N, Reese S, Ptak L, Aziz F, Parajuli S, Jucaud V, Denham S, Mishra A, Cascalho M, Platt JL, Hematti P, Djamali A. Ixazomib for Desensitization (IXADES) in Highly Sensitized Kidney Transplant Candidates: A Phase II Clinical Trial. Kidney360. 2023 Jun 1;4(6):e796-e808. doi: 10.34067/KID.0000000000000113. Epub 2023 Mar 23. PMID 36951387

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Started | 10
Completed | 7
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 40.8 [28.0 to 60.1]
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 2
  30-39 years | 4
  40-49 years | 2
  50-59 years | 1
  60-69 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
cPRA [Count of Participants; unit: Participants] — Calculated Panel of Reactive Antibodies (cPRA) which estimates the percentage of donors with whom a particular recipient would be incompatible.
  Participants
    81-85% | 1
    86-90% | 2
    91-95% | 0
    96-100% | 7
Cause of ESRD [Count of Participants; unit: Participants] — End-Stage Renal Disease (ESRD)
  Participants
    Congenital | 3
    Diabetes Mellitus (DM) | 2
    Glomerulonephritis (GN) | 1
    Alport's Syndrome | 1
    Polycystic Kidney Disease (PKD) | 1
    Systemic Lupus Erythematosus (SLE) | 1
    Focal segmental glomerulosclerosis (FSGS) | 1
Previous Treatment [Count of Participants; unit: Participants]
  Previous kidney transplant | 7
  2 previous kidney transplants | 2
  Previous kidney and pancreas transplant | 1
Interval of Previous Treatment [Mean (Full Range); unit: years] | 11.1 [5.0 to 18.8]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Ixazomib: Percentage of Participants With > 20 Percent Decline in Calculated Panel Reactive Antibody (cPRA)
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Number analyzed (Participants) | 10
Participants | 0

2. Primary Outcome: Efficacy of Ixazomib: Percentage of Participants Received Successful Kidney Transplantation Within 12 Months
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Number analyzed (Participants) | 10
Participants | 2

3. Secondary Outcome: Safety of Ixazomib as Assesses by Percentage of Participants With Cardiovascular Complications Within 12 Months
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Number analyzed (Participants) | 10
Participants | 2

4. Secondary Outcome: Safety of Ixazomib as Assesses by Percentage of Participants With Hematological Complications Within 12 Months
Description: Hematological complications include leucopenia, anemia, and thrombocytopenia
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Number analyzed (Participants) | 10
Participants | 2

5. Secondary Outcome: Safety of Ixazomib as Assesses by Percentage of Participants With Malignancies Within 12 Months
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Number analyzed (Participants) | 10
Participants | 0

6. Secondary Outcome: Safety of Ixazomib as Assesses by Percentage of Participants With Gastrointestinal Symptoms Within 12 Months
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Number analyzed (Participants) | 10
Participants | 5

7. Secondary Outcome: Safety of Ixazomib as Assesses by Percentage of Participants Caught Infection Within 12 Months
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Number analyzed (Participants) | 10
Participants | 5

8. Secondary Outcome: Safety of Ixazomib as Assesses by Percentage of Participants With Thrombocytopenia Within 12 Months
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Number analyzed (Participants) | 10
Participants | 0

9. Secondary Outcome: Safety of Ixazomib: as Assesses by Percentage of Participants With Distal Neuropathy Within 12 Months
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Number analyzed (Participants) | 10
Participants | 1

10. Other Pre Specified Outcome: Change in Circulating BAFF Levels as Assessed by BAFF ELISA Assay
Description: B cell activating factor belonging to the TNF family (BAFF) are members of the TNF ligand superfamily. Plasma BAFF ELISA assays can be performed in 2-3 hours. It can be used as a marker of disease activity in sensitized patients.
Time Frame: Baseline, 3 months
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Number analyzed (Participants) | 10
pg/ml
  Baseline | 126 [113 to 146]
  3 months | 160 [155 to 240]

11. Other Pre Specified Outcome: Change in Circulating APRIL Levels as Assessed by APRIL ELISA Assay
Description: B cell activating factor belonging to a proliferation-inducing ligand (APRIL) are members of the TNF ligand superfamily. Plasma APRIL ELISA assay can be performed in 2-3 hours. It can be used as a marker of disease activity in sensitized patients.
Time Frame: Baseline, 3 months
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Highly Sensitized Kidney Transplant Candidates
Number analyzed (Participants) | 10
pg/ml
  Baseline | 163 [134 to 198]
  3 months | 172 [151 to 219]

ADVERSE EVENTS:
Time Frame: up to 12 months
Arm/Group | Highly Sensitized Kidney Transplant Candidates
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Highly Sensitized Kidney Transplant Candidates (N=10)
Aortic valve disease (Cardiac disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (4)
Thromboembolic event (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Highly Sensitized Kidney Transplant Candidates (N=10)
Bacteremia (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Gum infection (Infections and infestations) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 2 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (9)
Headache (Nervous system disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (6)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT03213158/Prot_SAP_000.pdf